CLINICAL TRIAL: NCT00356343
Title: Strength Training Using NMES for Children With Cerebral Palsy
Brief Title: Strength Training Using Neuromuscular Electrical Stimulation For Children With Cerebral Palsy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Shriners Hospitals for Children (Other); University of Delaware (Other)
Responsible Party: Samuel C.K. Lee, University of DE/Shriners Hospitals for Children
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: R01HD043859 (NIH)
Record Dates: First submitted 2006-07-25; First posted 2006-07-26 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Spastic Diplegic Cerebral Palsy
Keywords: NMES; Cerebral Palsy; Spastic Diplegia; Electrical Stimulation; Children
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- NMES Strengthening Group (Experimental): Subjects will complete 12 weeks of NMES isometric strength training using implanted electrodes in bilateral quadriceps and triceps surae muscles.
  Interventions: Device: NMES Strength Training
- Control Group (No Intervention): No Intervention Control Group
- Volitional Strengthening (Active Comparator): Subjects will complete 12 weeks of volitional isometric strength training of bilateral quadriceps and triceps surae muscles.
  Interventions: Other: Volitional Strength Training

INTERVENTIONS:
Device: NMES Strength Training — Subjects will complete 12 weeks of NMES isometric strength training using implanted electrodes in bilateral quadriceps and triceps surae muscles.
  Arms: NMES Strengthening Group
Other: Volitional Strength Training — Subjects will complete 12 weeks of volitional isometric strength training of bilateral quadriceps and triceps surae muscles.
  Arms: Volitional Strengthening

SUMMARY:
The purpose of this study is to determine if using high-intensity, short-duration, intermittent neuromuscular electrical stimulation (NMES) is better than volitional exercise in increasing quadriceps femoris and triceps surae force-generating potential and gross motor function in children with cerebral palsy.

DETAILED DESCRIPTION:
The overall goal of this study is to determine if using high-intensity, short-duration, intermittent neuromuscular electrical stimulation (NMES) is better than volitional exercise in increasing quadriceps femoris and triceps surae force-generating potential and gross motor function in children with cerebral palsy. This study consists of a randomized controlled trial in which the effects of NMES applied to the quadriceps femoris and triceps surae are compared to the effects of volitional isometric exercise and a non-exercising control group. This project assesses the ability of NMES to increase muscle force generating ability, the mechanisms behind changes in force generating ability, and the effects of training on spatiotemporal parameters of gait and gross motor function in children with cerebral palsy.

Subjects is the NMES group will be implanted with percutaneous electrodes in the medial and lateral heads of the gastrocnemius and the quadriceps (3 electrodes in each lower extremity, implanted bilaterally). During the intervention phase, these subjects will undergo 15 electrically-elicited contractions in each of the implanted muscle groups three times/week (at home), while positioned on an exercise board to maintain good alignment and facilitate isometric contractions. Subjects in the volitional group will perform 15 isometric contractions in each muscle group (quadriceps, triceps surae), while positioned on an exercise board. The non-exercise control group will continue with typical activities, but no intervention will be administered. Subjects are assessed at baseline, 6 weeks into the intervention, 12 weeks into the intervention (at which point the intervention is withdrawn), and at a follow-up assessment 12 weeks after the withdrawal of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 7-12 years old
* Diagnosis of spastic diplegic cerebral palsy
* GMFCS level of II or III (able to walk indoors and outdoors with or without an assistive device)
* PROM requirements (<10 degree hip flexion contracture, >20 degrees of hip abduction, < 5 degrees of knee flexion contracture, > 45 degree popliteal angle, ankle dorsiflexion to neutral with knee extension)
* Sufficient cognitive/communication skills to perform volitional muscle contractions and complete data collection procedures

Exclusion Criteria:

* Significant orthopedic impairments (hip MIGR > 40%, significant scoliosis)
* Must be at least one year post orthopedic surgery
* Must be at least 6 months post botulinum toxin injections
* Uncontrolled seizure activity

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2004-07; Primary Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Force generating ability of quadriceps femoris and triceps surae (MVIC) | Pre, Mid, Post, Washout
Voluntary muscle activation during a Maximal Volitional Isometric Contraction (MVIC) | Pre, Mid, Post, Washout
Antagonist coactivation during an agonist MVIC | Pre, Mid, Post, Washout
Contractile properties as assessed via electrically-elicited tests | Pre, Mid, Post, Washout
Fatiguability of muscle as assessed via electrically-elicited tests | Pre, Mid, Post, Washout
Muscle cross-sectional area of quadriceps femoris and triceps surae (via MRI with fat suppression) | Pre, Mid, Post, Washout
Spatiotemporal parameters of gait | Pre, Mid, Post, Washout
Gross Motor Function Measure | Pre, Mid, Post, Washout
Timed Up and Go | Pre, Mid, Post, Washout
Parent and child report via questionnaires (PODCI, COPM) | Pre, Mid, Post, Washout

CONTACTS AND LOCATIONS:
Overall Officials: Samuel CK Lee, PhD, PT, Principal Investigator — University of Delaware, Shriners Hospitals for Children
Locations (1):
- Shriners Hospitals for Children, Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Stackhouse SK, Binder-Macleod SA, Lee SC. Voluntary muscle activation, contractile properties, and fatigability in children with and without cerebral palsy. Muscle Nerve. 2005 May;31(5):594-601. doi: 10.1002/mus.20302. PMID 15779003